CLINICAL TRIAL: NCT02121275
Title: Lung Ultrasound for the Detection of Pulmonary Atelectasis in the Perioperative Period
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Roman Ullrich, MD, Medical University of Vienna
Other Study IDs: LUS
Record Dates: First submitted 2014-04-02; First posted 2014-04-23 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Pulmonary Atelectases
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Laparoscopic surgery: Patients undergoing laparoscopic surgery under general anaesthesia, patients undergo ultrasound of the lungs and electric impedance tomography at 4 times during anaesthesia
  Interventions: Device: Ultrasound of the lungs; Device: Electric impedance tomography

INTERVENTIONS:
Device: Ultrasound of the lungs — Ultrasound examination of the lungs
  Other Names: Sonosite ultrasound device (M-Turbo)
Device: Electric impedance tomography — Electric impedance tomography (EIT) is a noninvasive tool based on the measurement of electrical impedance changes within the thorax and lung tissue during ventilation and depicts the regional changes in ventilation in real time. To use electric impedance tomography 16 electrodes are applied in a circular fashion around the patient's chest, typically at the level of the 7th intercostal space.
  Other Names: EIT (Pulmovista, Draeger)

SUMMARY:
Atelectases (collapsed lung areas) of 15-20% of total lung occur in up to 90% of patients who are anaesthetized and intubated. The goal of the present prospective study is to detect atelectatic areas in the perioperative period in the lungs of patients undergoing elective laparoscopic surgery non-invasively and without x-ray exposure. Results of lung ultrasound (LUS) as the experimental method will be compared to the results of Electrical Impedance Tomography (EIT) as the reference technique for the detection of atelectasis. A device for peripheral Oxygen saturation measurement (MASIMO Radical-8) will detect changes in ventilation. The investigators want to confirm or disprove former findings of the appearance of intraoperative atelectases and to prove that ultrasound is a valid tool for detection of atelectases.

ELIGIBILITY:
Inclusion Criteria:

* Male or female,
* age 18 - 75
* BMI < 30
* Laparoscopic operation

Exclusion Criteria:

* Pregnancy
* Pulmonary infection
* Chronic pulmonary diseases
* Morbid Obesity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective laparoscopic surgery at the Medical University of Vienna
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-09-06 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between evidence of atelectasis in lung ultrasound and evidence of atelectasis in electric impedance tomography | on the day of laparoscopic surgery, expected average 2 hours in total
  Measurements, requiring 5 minutes each, are performed before induction of anaesthesia, after intubation, immediately before extubation and immediately after extubation. Outcome measure: comparison of how often atelectases are detected by lung ultrasound (experimental method) versus by electric impedance tomography (standard method)

SECONDARY OUTCOMES:
respiratory variability of oxygen saturation | on the day of laparoscopic surgery, expected average 2 hours in total
  from induction of anaesthesia until extubation

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ullrich, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Dept. of Anesthesiology and General Intensive Care, Vienna, Austria